CLINICAL TRIAL: NCT00813696
Title: Gemcitabine vs Gemcitabine + Cisplatin in the Treatment of Advanced Pancreatic Cancer (Stage II III IV)
Brief Title: Gemcitabine or Gemcitabine and Cisplatin in the Treatment of Advanced Pancreatic Cancer
Acronym: GIP-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituti Tumori Giovanni Paolo II (Network)
Collaborators: Gruppo Oncologico Italia Meridionale (Other); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other); Gruppo Oncologico Italiano di Ricerca Clinica (Other); Cattedra di Endocrinochirurgia, Università di Verona (Unknown)
Responsible Party: Giuseppe Colucci, GOIM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIP-1
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Pancreatic Cancer
Keywords: chemotherapy; advanced cancer; inoperable; Stage II, III, IV
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): cisplatin + gemcitabine
  Interventions: Drug: gemcitabine; Drug: cisplatin
- B (Active Comparator): gemcitabine
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — 1000 mg/m2 IV weekly for 7 weeks. Starting at week 9, gemcitabine 1000 mg/m2 on days 1, 8, and 15 every 4 weeks
Drug: cisplatin — 25 mg/m2 IV on days 1, 8, and 15 every 4 weeks
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the impact of the addition of cisplatin to gemcitabine in the treatment of patients with inoperable advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis pancreatic cancer
* inoperable stage II or stage III or IV disease(UICC, 1997)
* Age 18 to 75 years
* Karnofsky Performance status > 50
* Signed informed consent

Exclusion Criteria:

* Previous chemotherapy
* Cerebral metastases
* Previous malignancies in past 5 years excluding adequately treated basal or spinocellular skin cancers and insitu cervical cancer
* Leukocytes < 4000 or neutrophils < 2000 or platelets < 100000 or hemoglobin < 10 g/dl
* Creatinine value > upper normal limit
* GOT or GPT > 2.5 times upper normal limit or bilirubin > 1.5 times upper normal limit in absence of hepatic metastases
* Congestive heart failure, severe cardiac arrhythmias or coronary ischemic disease
* Other concurrent disease that would, in the investigator's opinion, contraindicate the use of the study drugs
* Inability to provide informed consent
* Inability to comply with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-04; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
overall survival | 9 months

SECONDARY OUTCOMES:
clinical benefit response | baseline and at end of every cycle of therapy
quality of life | baseline and at end of every cycle of therapy
objective response | after 7 weeks of therapy
time to progression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Colucci, M.D., Principal Investigator — Istituto Tumori Giovanni Paolo II; Roberto Labianca, M.D., Principal Investigator — Ospedale Riuniti Bergamo; Francesco Di Costanzo, M.D., Principal Investigator — Azienda Ospedaliera Careggi; Stefano Cascinu, M.D., Principal Investigator — Ospedale Riuniti Umberto I-Lancise-Salese; Paolo Pederzoli, M.D., Principal Investigator — Policlinico G.B. Rossi, Verona; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples
Locations (45):
- Italy (45):
  - Ospedal Miulli, Acquaviva delle Fonti
  - Ospedale Regionale Torrette, Ancona
  - Presidio Osp. Alto Garda e Ledro, Arco
  - Centro Riferimento Oncologico, Aviano
  - Istituto Oncologico Giovanni Paolo II, Bari
  - Azienda Ospedaliera G. Rummo, Benevento
  - Ospedale Fatebenefratelli, Benevento
  - Ospedale Riuniti, Bergamo
  - Ospedale degli Infermi, Biella
  - Ospedale Regionale, Bolzano
  - Policlinico Universitario, Cagliari
  - Ospedale A. Cardarelli, Campobasso
  - Ospedale Ramazzini, Carpi
  - Centro Catanese di Oncologia, Catania
  - Università di Chieti "D'Annunzio", Chieti
  - Ospedale Valduce, Como
  - Ospedale Santa Croce, Fano
  - Azienda Ospedaliera Universitaria, Ferrara
  - Azienda Ospedale Careggi, Florence
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Ospedale Umberto I, Lugo
  - Pres. Osp. di Manerbio, Manerbio
  - Ospedale L. Sacco, Milan
  - Ospedale San Paolo, Milan
  - Ospedale G. Moscati, Monteforte Irpino
  - Ospedale San Gerardo, Monza
  - Istituto Nazionale Tumori, Napoli
  - Ospedale Cardarelli, Napoli
  - Ospedale Civile, Olbia
  - Casa di Cura La Maddalena, Palermo
  - Policlinico Giaccone, Palermo
  - Ospedale San Salvatore-Muraglia, Pesaro
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale San Carlo, Potenza
  - Azienda Policlinico S. Andrea, Roma
  - Ospedale Fatebenefratelli, Roma
  - Ospedale San Raffaele, Roma
  - Policlinico Militare Celio, Roma
  - Polo Oncologico Istituto Regina Elena, Roma
  - Ospedale Civile, Rovereto
  - Ospedale Civile, Rovigo
  - Centro Oncologico, S. Vito Al Tagliamento
  - Ospedale Santa Chiara, Trento
  - Azienda Ospedaliera Treviglio-Caravaggio, Treviglio
  - Ospedale San Bortolo, Vicenza

REFERENCES:
- [Derived] Colucci G, Labianca R, Di Costanzo F, Gebbia V, Carteni G, Massidda B, Dapretto E, Manzione L, Piazza E, Sannicolo M, Ciaparrone M, Cavanna L, Giuliani F, Maiello E, Testa A, Pederzoli P, Falconi M, Gallo C, Di Maio M, Perrone F; Gruppo Oncologico Italia Meridionale (GOIM); Gruppo Italiano per lo Studio dei Carcinomi dell'Apparato Digerente (GISCAD); Gruppo Oncologico Italiano di Ricerca Clinica (GOIRC). Randomized phase III trial of gemcitabine plus cisplatin compared with single-agent gemcitabine as first-line treatment of patients with advanced pancreatic cancer: the GIP-1 study. J Clin Oncol. 2010 Apr 1;28(10):1645-51. doi: 10.1200/JCO.2009.25.4433. Epub 2010 Mar 1. PMID 20194854